CLINICAL TRIAL: NCT03303300
Title: The Five-repetition Sit-to-stand Test as an Objective Measure of Functional Impairment in Patients With Lower Back Pain or Radiculopathy
Brief Title: The Five-repetition Sit-to-stand Test for Lower Back Pain or Radiculopathy
Acronym: 5R-STS
Status: Completed | Type: Observational
Sponsor: Marc Schröder (Other)
Responsible Party: Sponsor-Investigator, Marc Schröder, MD, PhD, Bergman Clinics
Organization: Bergman Clinics (Other)
Other Study IDs: 5RSTS
Record Dates: First submitted 2017-09-23; First posted 2017-10-06 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Herniated Disc; Stenosis, Spinal; Nerve Root Compress;Lumbosac
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The five-repetition sit-to-stand test (5R-STS) has been used in many medical disciplines, but has never been correlated with or validated in regard to degenerative spinal diseases. The investigators aim to assess the possibility of using the standardized 5R-STS as an objective measure of functional impairment and pain severity in patients with degenerative lumbar spinal diseases.

ELIGIBILITY:
This study will include 100 Patients:

Inclusion Criteria:

* Degenerative diseases of the lumbar spine (Herniated disc, lumbar stenosis, spondylolisthesis, degenerative disc disease)
* Symptoms of lower back pain, neurogenic claudication, or radiculopathy

Exclusion Criteria:

* Hip or Knee prosthetics
* Walking aides

This study will also include 25 healthy volunteers:

Inclusion Criteria:

- No degenerative spinal or lower extremity complaints

Exclusion Criteria:

* Back pain, leg pain, other lower extremity-related complaints
* Knee or hip prosthetics
* Walking aides

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients with degenerative lumbar spinal diseases that are seen in outpatient consultations will be recruited. All tests and questionnaires are part of the normal clinical assessment of the study center; The patients are thus not required to make any extra efforts.
  25 healthy volunteers (the authors and volunteers from the department) will be included to get baseline data for the 5R-STS in healthy people
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-03 (Actual)

PRIMARY OUTCOMES:
5R-STS | 0 weeks
  The result of the standardized 5R-STS in seconds. If the patient is unable to complete the test, the results is noted as "not possible".

SECONDARY OUTCOMES:
VAS back pain | 0 weeks
  Validated questionnaire (VAS BP) will be used to correlate the 5R-STS results with validated measures of functional impairment and pain severity.
VAS leg pain | 0 weeks
  Validated questionnaire (VAS LP) will be used to correlate the 5R-STS results with validated measures of functional impairment and pain severity.
EQ-5D-3L | 0 weeks
  Validated questionnaire (EQ-5D-3L) will be used to correlate the 5R-STS results with validated measures of functional impairment and pain severity.
Oswestry Disability Index | 0 weeks
  Validated questionnaire (ODI) will be used to correlate the 5R-STS results with validated measures of functional impairment and pain severity.
Roland-Morris-Disability Questionnaire | 0 weeks
  Validated questionnaire (RMDBQ) will be used to correlate the 5R-STS results with validated measures of functional impairment and pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Bergman Clinics, Naarden, Netherlands

REFERENCES:
- [Derived] Klukowska AM, Staartjes VE, Vandertop WP, Schroder ML. Predictors of five-repetition sit-to-stand test performance in patients with lumbar degenerative disease. Acta Neurochir (Wien). 2023 Jan;165(1):107-115. doi: 10.1007/s00701-022-05441-1. Epub 2022 Dec 7. PMID 36477416
- [Derived] Staartjes VE, Klukowska AM, Schroder ML. Association of maximum back and leg pain severity with objective functional impairment as assessed by five-repetition sit-to-stand testing: analysis of two prospective studies. Neurosurg Rev. 2020 Oct;43(5):1331-1338. doi: 10.1007/s10143-019-01168-3. Epub 2019 Aug 26. PMID 31451936
- [Derived] Staartjes VE, Schroder ML. The five-repetition sit-to-stand test: evaluation of a simple and objective tool for the assessment of degenerative pathologies of the lumbar spine. J Neurosurg Spine. 2018 Oct;29(4):380-387. doi: 10.3171/2018.2.SPINE171416. Epub 2018 Jun 29. PMID 29957147